CLINICAL TRIAL: NCT06088654
Title: A Phase 1/2, Open-Label, Multicenter Trial Investigating the Safety, Tolerability, and Preliminary Antineoplastic Activity of IPH6501 in Patients With Relapsed and/or Refractory CD20-expressing Non-Hodgkin Lymphoma
Brief Title: Phase1/2 Study of IPH6501 in Patients With Relapsed /Refractory B-Cell Non-Hodgkin Lymphoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Innate Pharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IPH6501-101
Record Dates: First submitted 2023-10-12; First posted 2023-10-18 (Actual); Last update posted 2025-04-02 (Actual); Status verified 2025-03

CONDITIONS: Non Hodgkin Lymphoma
Keywords: ANKET®; NK cell engager; tetraspecific NK cell engager
MeSH Terms: conditions — Lymphoma, Non-Hodgkin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- IPH6501 monotherapy (Experimental)
  Interventions: Drug: IPH6501

INTERVENTIONS:
Drug: IPH6501 — phase 1 (dose finding) and phase 2 (dose expansion)

SUMMARY:
This is an international, first-in-human, multicenter, open-label Phase 1/2 study to evaluate the safety profile, tolerability of IPH6501, and determine the recommended phase 2 dose (RP2D) for patients with B-Cell non-Hodgkin lymphoma.

DETAILED DESCRIPTION:
In Phase 1 - Dose finding, patients with advanced histologically confirmed, documented CD20+ B-cell non-Hodgkin lymphoma (NHL) will be enrolled. The dose finding part will include 2 sub-parts: Dose escalation will determine the Maximum Tolerated Dose (MTD) or the highest tested dose, Dose assessment will determine RP2D.

In Phase 2 - Dose expansion, one or more cohorts will be selected with patients with subtypes of advanced histologically confirmed, documented CD20+ B-cell non-Hodgkin lymphoma.

ELIGIBILITY:
Main Inclusion criteria

* Patients with advanced histologically confirmed, documented CD20+ B-cell non-Hodgkin's lymphoma (NHL) including the following types defined by WHO 2016: Diffuse Large B Cell Lymphoma (DLBCL); high grade; thymic; Follicular Lymphoma (FL); Mantle cell lymphoma (MCL); Marginal zone lymphoma (MZL)
* Relapsed, progressive and/or refractory disease without established alternative therapy
* Must have received at least 2 prior systemic therapies including at a minimum anti-CD20 antibody therapy (e.g., rituximab) potentially in combination with chemotherapy and/or relapsed after autologous stem cell rescue.
* Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 2
* Adequate organ and hematological function
* Able to provide a fresh biopsy from a safely accessible site (or historical biopsy), per investigator determination.

Main Exclusion Criteria

* Patients with another invasive malignancy in the last 2 years
* Prior chemotherapy, immunotherapy or other anti-cancer therapy within less than 4 weeks before study drug administration.
* Autologous stem cell transplant or treatment with CAR-T (Chimeric Antigen Receptor T-Cell) cell therapy within 100 days prior to first dose of study drug
* Subjects with brain or subdural metastases are not eligible, nor those with history of central nervous system (CNS) lymphoma
* Current or past history of CNS disease, such as stroke, epilepsy, CNS vasculitis, or neurodegenerative disease.
* Known history of infection with human immunodeficiency virus (HIV) or hepatitis B or C
* Major surgery within 4 weeks before the first dose of study drug
* Comorbidities including diabetes, cardiovascular diseases, immunodeficiencies/autoimmune condition
* Pregnant / breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 184 (Estimated)
Dates: Start 2024-03-04 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Safety and tolerability | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To evaluate the safety profile (including dose limiting toxicities (DLT(s), the maximum tolerated dose (MTD) or highest tested dose), tolerability and determine the recommended phase 2 dose (RP2D)

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To investigate any preliminary antitumor activity
Duration Of Response (DoR) | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To investigate any preliminary antitumor activity
Progression Free Survival (PFS) | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To investigate any preliminary antitumor activity
Maximum Observed Plasma Concentration (Cmax) | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To characterize and evaluate the pharmacokinetic profile of IPH6501
Area Under the Plasma Concentration (AUC) | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To characterize and evaluate the pharmacokinetic profile of IPH6501
Incidence of antidrug antibodies (ADA) against IPH6501 | From time of informed consent through treatment period and including the follow-up: up to 22 months
  To evaluate the immunogenicity of IPH6501

CONTACTS AND LOCATIONS:
Locations (14):
- United States (5):
  - City of Hope, Duarte, California
  - Cedars Sinai, Los Angeles, California
  - Siteman Cancer Center, St Louis, Missouri
  - Icahn School Of Medicine At Mount Sinai, New York, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
- Australia (4):
  - Wollongong Private Hospital, Wollongong, New South Wales
  - Monash Health, Clayton, Victoria
  - Peninsula Private Hospital, Frankston, Victoria
  - Austin Health, Heidelberg
- France (5):
  - Institute Bergonie, Bordeaux
  - Centre Hospitalier Regional Universitaire de Lille, Lille
  - Hospices Civils de Lyon, Lyon
  - Hôpital de la Coception, Marseille
  - Centre Hospitalier Universitaire de Nantes, Nantes

IPD SHARING:
Plan to Share IPD: No